CLINICAL TRIAL: NCT02233933
Title: Randomized Trial of Argon Plasma Coagulation Versus Argon Plasma Coagulation and Hemospray in the Therapy of Radiation Proctitis
Brief Title: Trial of Argon Plasma Coagulation Versus APC and APC and Hemospray in the Treatment of Radiation Proctitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Alan Weiss, Principal Investgator, British Columbia Cancer Agency
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RadP
Record Dates: First submitted 2014-08-28; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Rectal Bleeding
Keywords: radiation proctitis; bleeding; therapy
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhage | interventions — hemospray

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- argon plasma coagulation (Active Comparator): argon plasma coagulation of radiation proctitis
  Interventions: Other: Hemospray
- argon plasma coagulator and hemospray (Experimental): treatment of radiation proctitis with argon plasma coagulator followed by application of hemospray
  Interventions: Other: Hemospray

INTERVENTIONS:
Other: Hemospray — hemospray is used after argon coagulation to stop bleeding

SUMMARY:
Randomized trial of Argon Plasma Coagulation compared with Argon Plasma Coagulation and Hemospray in the therapy of bleeding from Radiation Proctitis

DETAILED DESCRIPTION:
20 patients with Radiation Proctitis will be randomized to receive either Argon Plasma Coagulation therapy alone or therapy with APC followed by Hemospray administration ;the treatment in each arm is administered during a sigmoidoscopic examination

ELIGIBILITY:
Inclusion Criteria:

* bleeding from radiation proctitis

Exclusion Criteria:

* pregnancy bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
cessation of rectal bleeding | 12 months
  treatment of one group of patients with Radiation Proctitis with Argon Plasma Coagulator ( APC) and a second group will be treated with APC and Hemospray

SECONDARY OUTCOMES:
number of treatments required to achieve cessation of rectal bleeding | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan A Weiss, MD, Principal Investigator — BCCA
Locations (1):
- British Columbia Cancer Clinic, Vancouver, British Columbia, Canada